CLINICAL TRIAL: NCT00441857
Title: The Effect of Three Different Stanol Ester Doses in Margarines on Cholesterol Absorption Efficiency
Brief Title: Effect of Plant Stanols on Cholesterol Absorption
Acronym: DOSE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Oy Foodfiles Ltd (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DOSE
Record Dates: First submitted 2007-02-28; First posted 2007-03-01 (Estimated); Last update posted 2007-07-06 (Estimated); Status verified 2007-07

CONDITIONS: Hypercholesterolemia
Keywords: plant sterols; plant stanols; cholesterol absorption
MeSH Terms: conditions — Hypercholesterolemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: plant stanol consumption

SUMMARY:
This study aims to measure the effect of three different doses of plant stanols in margarine on the cholesterol absorption efficiency in subjects with mildly to moderately increased serum LDL cholesterol concentrations

DETAILED DESCRIPTION:
Serum cholesterol lowering effect of plant sterols is well established and it is also known that plant stanols inhibit the absorption of cholesterol. However, there is lack of dose-response studies directly measuring the cholesterol absorption efficiency during prolonged consumption of plant stanols. Therefore this study aims to measure the cholesterol absorption efficiency at different plant stanol consumption levels using a stable isotope tracer method.

Subjects will be randomized in their study groups that consume 20 g of margarine with different doses of plants stanols (0.8, 1.6 and 2.0g) based on cholesterol absorption efficiency at screening (high and low absorbers randomised separately). Cholesterol absorption test with cholesterol tracer will be conducted twice: at baseline and after 2-3 weeks margarine consumption period.

Cholesterol absorption efficiency will also be examined by indirect method i.e. by following the concentrations of serum cholesterol precursors and plant sterols in blood. In addition serum total, LDL and HDL cholesterol and triglycerides are followed.

ELIGIBILITY:
Inclusion Criteria:

* healthy adults with mild to moderate hypercholesterolemia

Exclusion Criteria:

* lipid lowering medication
* pregnancy or lactation
* severe diseases (inc. diabetes, unstable CVD, malignant diseases)
* severe obesity
* regular plant sterol consumption

Ages: 25 Years to 68 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60
Dates: Start 2007-03; Study Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
cholesterol absorption efficiency

SECONDARY OUTCOMES:
changes in blood lipids

CONTACTS AND LOCATIONS:
Overall Officials: Sakari A Nieminen, MD, Principal Investigator — Oy Foodfiles Ltd
Locations (1):
- Oy Foodfiles Ltd, Kuopio, Finland